CLINICAL TRIAL: NCT05598658
Title: Effect of Remote Ischemic Conditioning on Cerebral Hemodynamics in Patients After Intravenous Thrombolysis (RICCH-IVT)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yi Yang (Other)
Responsible Party: Sponsor-Investigator, Yi Yang, Associated Dean of First Hospital of Jilin University, The First Hospital of Jilin University
Organization: The First Hospital of Jilin University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RICCH-IVT
Record Dates: First submitted 2022-10-25; First posted 2022-10-28 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Remote Ischemic Conditioning
Keywords: Remote Ischemic Conditioning; Intravenous Thrombolysis; Cerebral Hemodynamics; Cerebral Autoregulation; Cerebral Blood Flow Velocity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RIC group (Active Comparator): Remote ischemic conditioning (RIC) is induced by 4 cycles of 5 min of healthy upper limb ischemia followed by 5 min re-perfusion. Limb ischemia was induced by inflation of a blood pressure cuff to 200 mm Hg. RIC will be conducted at 6 and 18-24 hours after intravenous thrombolysis.
  Interventions: Procedure: Remote ischemic conditioning
- Sham-RIC group (Placebo Comparator): Remote ischemic conditioning (RIC) is induced by 4 cycles of 5 min of healthy upper limb ischemia followed by 5 min re-perfusion. Limb ischemia was induced by inflation of a blood pressure cuff to 60 mm Hg. RIC will be conducted at 6 and 18-24 hours after intravenous thrombolysis.
  Interventions: Procedure: Sham remote ischemic conditioning

INTERVENTIONS:
Procedure: Remote ischemic conditioning — Remote ischemic conditioning (RIC) is induced by 4 cycles of 5 min of healthy upper limb ischemia followed by 5 min reperfusion. Limb ischemia was induced by inflations of a blood pressure cuff to 200 mm Hg.
  Arms: RIC group
Procedure: Sham remote ischemic conditioning — Sham remote ischemic conditioning (RIC) is induced by 4 cycles of 5 min of healthy upper limb ischemia followed by 5 min reperfusion. Limb ischemia was induced by inflations of a blood pressure cuff to 60 mm Hg.
  Arms: Sham-RIC group

SUMMARY:
The purpose of this study is to determine the effect of remote ischemic conditioning on cerebral hemodynamics in patients after intravenous thrombolysis

DETAILED DESCRIPTION:
In this study, cases of ischemic stroke who undergo intravenous thrombolysis within 4.5 hours from onset are included. The RIC group receive basic treatment and remote ischemic conditioning for 200mmHg at 6 and 18-24 hours after intravenous thrombolysis. The sham-RIC group receive basic treatment and remote ischemic conditioning for 60mmHg at 6 and 18-24 hours after intravenous thrombolysis. Both groups underwent cerebral hemodynamics after RIC and recorded the relevant indexes. The investigators aimed to determine the effect of remote ischemic conditioning on cerebral hemodynamics in patients after intravenous thrombolysis.

ELIGIBILITY:
Inclusion Criteria:

1. age ≥ 18 and < 80 years, both sexes;
2. a clear clinical diagnosis of acute ischemic stroke and treatment with standard rt-PA (0.9 mg/kg) IVT within 4.5 h of stroke onset;
3. pre-onset modified Rankin Scale (mRS) score ≤1;
4. baseline National Institute of Health Stroke Scale (NIHSS) score ≥5 and ≤25;
5. Glasgow Coma Scale score ≥8.

Exclusion Criteria:

1. having received bridging therapy (IVT plus mechanical thrombectomy);
2. previous history of atrial fibrillation or electrocardiographic evidence of atrial fibrillation;
3. contraindications to RIC treatment or previous RIC treatment or similar treatment;
4. pregnancy or breastfeeding;
5. life expectancy of ≤3 months or inability to complete the study for other reasons;
6. unwillingness to be followed up or poor treatment compliance or participation in other clinical studies;
7. had insufficient bilateral temporal bone windows for insonation of the middle cerebral artery.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-01-12 (Actual); Study Completion 2024-04-12 (Actual)

PRIMARY OUTCOMES:
Cerebral autoregulation parameter | 1-10 days
  Cerebral autoregulation parameters derived from transfer function analysis. Continuous cerebral blood flow velocities of bilateral middle cerebral artery will be assessed noninvasively using transcranial Doppler. Spontaneous arterial blood pressure will be simultaneously recorded using a servo-controlled plethysmograph on the left or right middle finger with an appropriate finger cuff size. Transfer function analysis will be used to derive the autoregulatory parameter.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Hospital of Jilin University, Changchun, Jilin, China